CLINICAL TRIAL: NCT02531308
Title: A Phase ll Study Evaluating the Efficacy and Safety of Metformin in Combination With Standard Induction Therapy (RM-CHOP) for Previously Untreated Aggressive Diffuse Large B-cell Lymphoma
Brief Title: Metformin in Combination With Standard Induction Therapy for Large B-cell Lymphoma (DLBCL)
Acronym: DLBCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYM2014-MET-R-CHOP | 15100503
Record Dates: First submitted 2015-07-27; First posted 2015-08-24 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: diffuse large b-cell lymphoma (DLBCL),; lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Lymphoma | interventions — Metformin; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CHOP with Metformin (Experimental): Rituximab 375 mg/m2 IV infusion Day 1 Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Vincristine 1.4 mg/m2 (2 mg cap) IV Day 1 Prednisone 100 mg PO Days 1-5 Pegfilgrastim 6 mg subcutaneous within 72 hours of cyclophosphomide Metformin 500 mg PO daily D 1-7, 500 mg twice daily D8-21, 850 mg twice daily D22 - 30days post study.
  Cycles are 21 days. Above treatment given for 4 cycles, then restaging done. If complete response (CR) or partial response (PR), 2 more cycle given; stable disease (SD) or progressive disease (PD)- salvage therapy off study.
  Interventions: Drug: Metformin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: pegfilgrastim

INTERVENTIONS:
Drug: Metformin — Metformin upregulates AMPK activity which has been shown to have an anti-proliferative effect on lymphoma cells.
  Other Names: Glucophage, Glucophage XR, Glumetza, Fortamet, Riomet.
Drug: Rituximab — monoclonal antibody against protein CD20 primarily found on the surface of B-cells
  Other Names: Rituxan, Zytux, Mab thera
Drug: Cyclophosphamide — Interferes with DNA replication
  Other Names: Endoxan, Cytoxan, Neosar, Procytox, Revimmune, Cycloblastin
Drug: Doxorubicin — anthracycline antitumor antibiotic
  Other Names: Adriamycin
Drug: Vincristine — Inhibits cell mitosis causing cell death.
  Other Names: Oncovin
Drug: Prednisone — a synthetic corticosteroid drug that is particularly effective as an immunosuppressant drug. It is used to treat certain inflammatory diseases
  Other Names: Deltasone
Drug: pegfilgrastim — stimulates the level of white blood cells (neutrophils).
  Other Names: Neulasta

SUMMARY:
Evaluation of impact of metformin on 2 year progression-free survival (PFS) rate in subjects with previously untreated DLBCL when added to standard induction therapy. (R-CHOP)

DETAILED DESCRIPTION:
Newly diagnosed histologically confirmed CD20 positive previously untreated diffuse large B-cell lymphoma to receive up to 4-6 cycles (21 day cycles) of:

R-CHOP: Rituximab 375 mg/m2 IV infusion Day 1 Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Vincristine 1.4 mg/m2 IV Day 1 (cap @ 2mg) Prednisone 100mg PO daily Days 1-5 Pegfilgrastim 6 mg subcutaneously within 72 if start if cycle Metformin 500 mg PO daily Cycle 1 Days 1-7 Metformin 500 mg PO twice daily Cycle 1 Days 7-21 Metformin 850 mg PO twice daily starting on day 22 and and continuing throughout remainder of cycles plus 22 days post treatment.

Restaging will be done after the 4th cycle is complete. Subjects will be monitored with labs and physical exams throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Diffuse Large B-cell Lymphoma (DLBCL) as documented by medical records and with histology based on criteria established by the World Health Organization

   a. subtyping is required for DLBCL
2. No prior therapy for diagnosis of DLBCL
3. Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of equal to or greater than 1 lesion that measures >1.5 cm in the longest diameter and > 1.0 cm in the longest perpendicular diameter assessed by CT or MRI) or bone marrow involvement
4. Eastern Cooperative Oncology Group performance score of 0-2
5. Life expectancy of at least 6 months
6. No history of medication dependent diabetes mellitus
7. Required screening laboratory data (within 4 weeks prior to start of study drug) -

Exclusion Criteria:

1. Patients already on any class of anti-diabetic medication including metformin, insulin analogues, sulfonylureas, thiazolidinediones (TZDs) and the incretin-based therapies or clear need for therapeutic intervention based on fasting blood glucose
2. Known histological transformation from indolent non-Hodgkins Lymphoma (NHL) or chronic lymphocytic leukemia (CLL) to an aggressive form of NHL (ie, Richter transformation)
3. Double or triple hit lymphomas
4. Known active cent4ral nervous system or leptomeningeal lymphoma
5. Presence of known intermediate or high-grade myelodysplastic syndrome
6. History of a non-lymphoid malignancy within the last 3 years (see protocol for exceptions)
7. Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of start of study
8. Ongoing, drug-induced liver injury, chronic active Hepatitis C Virus (HCV), chronic active Hepatitis B Virus (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
9. HIV positive
10. Ongoing inflammatory bowel disease
11. Ongoing alcohol or drug addiction
12. Pregnancy
13. History of prior allogeneic bone marrow progenitor cell or solid organ transplantation.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reem Karmali, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- R-CHOP With Metformin: Rituximab 375 mg/m2 IV infusion Day 1 Cyclophosphamide 750 mg/m2 IV Day 1 Doxorubicin 50 mg/m2 IV Day 1 Vincristine 1.4 mg/m2 (2 mg cap) IV Day 1 Prednisone 100 mg PO Days 1-5 Pegfilgrastim 6 mg subcutaneous within 72 hours of cyclophosphomide Metformin 500 mg PO daily D 1-7, 500 mg twice daily D8-21, 850 mg twice daily D22 - 30days post study.
  Cycles are 21 days. Above treatment given for 4 cycles, then restaging done. If complete response (CR) or partial response (PR), 2 more cycle given; stable disease (SD) or progressive disease (PD)- salvage therapy off study.
  Metformin: Metformin upregulates AMPK activity which has been shown to have an anti-proliferative effect on lymphoma cells.
  Rituximab: monoclonal antibody against protein CD20
  Cyclophosphamide: Interferes with DNA replication
  Doxorubicin: anthracycline antitumor antibiotic
  Vincristine: Inhibits cell mitosis causing cell death.
  Prednisone: a synthetic cortic
Period: Overall Study
Arm/Group | R-CHOP With Metformin
Started | 5
Completed | 2
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | R-CHOP With Metformin
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: rate of progression in patients 2 years after diagnosis
Time Frame: 2 year
Population: The primary endpoint (2 year PFS rate) could not be determined as study was terminated prematurely prior to subjects reaching this milestone with confidentiality of concern for reporting collected data.
Arm/Group | R-CHOP With Metformin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | R-CHOP With Metformin
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-CHOP With Metformin (N=5)
Fever with urosepsis (Infections and infestations) | 1 (2) — 2 hospitalizations for above SAE
Pulmonary Embolism and DVT (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-CHOP With Metformin (N=5)
fatigue (General disorders) | 5 (5)
hypoglycemia (Endocrine disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 4
thrombocytopenia (Blood and lymphatic system disorders) | 2
neutropenia (Blood and lymphatic system disorders) | 3
cardiomyopathy (Cardiac disorders) | 2

LIMITATIONS AND CAVEATS:
Unable to report on endpoint of 2 year PFS as trial prematurely terminated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes